CLINICAL TRIAL: NCT05845489
Title: Efficacy and Safety of Clopidogrel for Primary Prevention in Patients With Subclinical Coronary Atherosclerosis Identified on Imaging
Brief Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Stenosis- CloPidogREl for Primary preVENTION (HOST-PREVENTION)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samjin Pharmaceutical Co., Ltd. (Industry); CKD Pharmaceutical Limited (Unknown); Hanmi Pharmaceutical co., ltd. (Other); Yuhan Pharmaceutical Company (Unknown); Daewoong Pharmaceutical Co. LTD. (Industry); Dong-A ST Co., Ltd. (Industry); IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-2212-044-1385
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; clopidogrel; prevention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel treatment group (Experimental): Patients assigned to the clopidogrel treatment group will maintain clopidogrel 75mg once a day for at least 5 years.
  Interventions: Drug: Clopidogrel treatment group
- No antiplatelet or anticoagulant group (Active Comparator): Patients assigned to the no antiplatelet or anticoagulant group will not prescribe antithrombotics for at least 5 years. However, when there is a medical need for antithrombotic therapy during the follow-up, the prescription of antithrombotics is permitted with reporting to the research board.
  Interventions: Other: No antiplatelet or anticoagulant group

INTERVENTIONS:
Drug: Clopidogrel treatment group — Patients assigned to the clopidogrel treatment group will maintain clopidogrel 75mg once a day for at least 5 years.
  Arms: Clopidogrel treatment group
Other: No antiplatelet or anticoagulant group — Patients assigned to the no antiplatelet or anticoagulant group will not prescribe antithrombotics for at least 5 years. However, when there is a medical need for antithrombotic therapy during the follow-up, the prescription of antithrombotics is permitted with reporting to the research board.
  Arms: No antiplatelet or anticoagulant group

SUMMARY:
The investigators will evaluate the efficacy and safety of clopidogrel for primary prevention in patients diagnosed with coronary atherosclerosis on imaging that did not require revascularization therapy.

The trial will test the hypothesis that clopidogrel is beneficial in preventing major adverse cardiovascular and cerebrovascular events (MACCE) in patients with subclinical coronary atherosclerosis identified on imaging.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most prevalent and lethal disease worldwide. Even though various studies have been performed regarding the prevention or treatment of CAD and its related cardiovascular events, the prevalence of CAD and the incidence of cardiovascular events are increasing.

Antiplatelet agents are among the most widely used drugs for preventing cardiovascular events. The efficacy of antiplatelet agents has been extensively proven in secondary prevention for cardiovascular events in CAD patients, and their use has been recommended in current guidelines. However, there is still controversy surrounding the prescription of antiplatelet agents for the primary prevention of cardiovascular events in CAD patients due to their unknown clear efficacy and risk of bleeding complications.

Recent studies reported the limited efficacy of aspirin in old patients, diabetes patients, or patients with cardiovascular events risks. However, the efficacy or safety of antiplatelet therapy in patients with subclinical coronary atherosclerosis has not been thoroughly investigated. These patients are at higher risk of cardiac death or myocardial infarction compared to patients without coronary atherosclerosis.

In this regard, the investigators will evaluate the efficacy and safety of clopidogrel for primary prevention in patients diagnosed with coronary atherosclerosis on imaging that did not require revascularization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥40 years
* Patients with subclinical coronary atherosclerosis identified from coronary CT angiography or coronary angiography within 2 years without clinical events after an imaging study
* Without significant coronary artery stenosis (Diameter stenosis >50%), which needs revascularization
* Agreement to give written informed consent

Exclusion Criteria:

* A history of a diagnosed cardiovascular or cerebrovascular disease (Type1 myocardial infarction, heart failure, peripheral artery disease, stroke, transient ischemic attack, carotid artery stenosis>50%, carotid artery intervention)
* A history of coronary artery intervention or coronary artery bypass graft surgery, which needs chronic maintenance of antiplatelet therapy
* Absolute contraindication or allergy to clopidogrel
* Patients receiving anticoagulants for other comorbidities
* A history of Bleeding diathesis, known coagulopathy, or major bleeding, BARC class ≥3, resulting in the stop of antiplatelet agents
* Planned surgery or intervention which needs to stop antiplatelet agents ≥1 month
* Presence of non-cardiac comorbidity with life expectancy ≤ 5 years at randomization
* Females with pregnancy or breast-feeding
* Patients who are thought to be inappropriate for the trial based on physicians' decision

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11086 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | at 2 years after the last enrollment
  A composite of all-cause death, non-fatal myocardial infarction, any coronary revascularization, ischemic stroke, or transient ischemic attack

SECONDARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | at 5 years after the last enrollment
  A composite of all-cause death, non-fatal myocardial infarction, any coronary revascularization, ischemic stroke, or transient ischemic attack
Net adverse clinical event | at 2 years and 5 years after the last enrollment
  A composite of all-cause death, non-fatal myocardial infarction, any coronary revascularization, ischemic stroke or transient ischemic attack, major bleeding
All-cause death | at 2 years and 5 years after the last enrollment
Non-fatal myocardial infarction | at 2 years and 5 years after the last enrollment
Any coronary revascularization | at 2 years and 5 years after the last enrollment
Ischemic stroke or Transient ischemic attack | at 2 years and 5 years after the last enrollment
Any non-coronary revascularization | at 2 years and 5 years after the last enrollment
Major bleeding events | at 2 years and 5 years after the last enrollment
  BARC classification, type 3 or 5
BARC type 2 bleeding events | at 2 years and 5 years after the last enrollment
BARC type 3 bleeding events | at 2 years and 5 years after the last enrollment
BARC type 5 bleeding events | at 2 years and 5 years after the last enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (54):
- South Korea (54):
  - Seoul National University Hospital, Seoul, Other
  - Andong Hospital, Andong
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do
  - Eulji University Hospital, Uijeongbu, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Myongji Hospital, Gyeonggi-do
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do
  - Sejong General Hospital, Bucheon, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Gyeonggi-do
  - Yonsei University Yongin Severance Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun
  - Catholic Kwandong University International St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
  - Jesus Hospital, Jeonju, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Pohang Stroke And Spine Hospital, Pohang
  - Chungnam National University Sejong Hospital, Sejong
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Seoul Hospital, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Veterans Health Service Medical Center, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yazdanyar A, Newman AB. The burden of cardiovascular disease in the elderly: morbidity, mortality, and costs. Clin Geriatr Med. 2009 Nov;25(4):563-77, vii. doi: 10.1016/j.cger.2009.07.007. PMID 19944261
- [Background] Hennekens CH, Dyken ML, Fuster V. Aspirin as a therapeutic agent in cardiovascular disease: a statement for healthcare professionals from the American Heart Association. Circulation. 1997 Oct 21;96(8):2751-3. doi: 10.1161/01.cir.96.8.2751. No abstract available. PMID 9355934
- [Background] Ajani UA, Ford ES, Greenland KJ, Giles WH, Mokdad AH. Aspirin use among U.S. adults: Behavioral Risk Factor Surveillance System. Am J Prev Med. 2006 Jan;30(1):74-7. doi: 10.1016/j.amepre.2005.08.042. PMID 16414427
- [Background] Ittaman SV, VanWormer JJ, Rezkalla SH. The role of aspirin in the prevention of cardiovascular disease. Clin Med Res. 2014 Dec;12(3-4):147-54. doi: 10.3121/cmr.2013.1197. Epub 2014 Feb 26. PMID 24573704
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] McNeil JJ, Wolfe R, Woods RL, Tonkin AM, Donnan GA, Nelson MR, Reid CM, Lockery JE, Kirpach B, Storey E, Shah RC, Williamson JD, Margolis KL, Ernst ME, Abhayaratna WP, Stocks N, Fitzgerald SM, Orchard SG, Trevaks RE, Beilin LJ, Johnston CI, Ryan J, Radziszewska B, Jelinek M, Malik M, Eaton CB, Brauer D, Cloud G, Wood EM, Mahady SE, Satterfield S, Grimm R, Murray AM; ASPREE Investigator Group. Effect of Aspirin on Cardiovascular Events and Bleeding in the Healthy Elderly. N Engl J Med. 2018 Oct 18;379(16):1509-1518. doi: 10.1056/NEJMoa1805819. Epub 2018 Sep 16. PMID 30221597
- [Background] ASCEND Study Collaborative Group; Bowman L, Mafham M, Wallendszus K, Stevens W, Buck G, Barton J, Murphy K, Aung T, Haynes R, Cox J, Murawska A, Young A, Lay M, Chen F, Sammons E, Waters E, Adler A, Bodansky J, Farmer A, McPherson R, Neil A, Simpson D, Peto R, Baigent C, Collins R, Parish S, Armitage J. Effects of Aspirin for Primary Prevention in Persons with Diabetes Mellitus. N Engl J Med. 2018 Oct 18;379(16):1529-1539. doi: 10.1056/NEJMoa1804988. Epub 2018 Aug 26. PMID 30146931
- [Background] Gaziano JM, Brotons C, Coppolecchia R, Cricelli C, Darius H, Gorelick PB, Howard G, Pearson TA, Rothwell PM, Ruilope LM, Tendera M, Tognoni G; ARRIVE Executive Committee. Use of aspirin to reduce risk of initial vascular events in patients at moderate risk of cardiovascular disease (ARRIVE): a randomised, double-blind, placebo-controlled trial. Lancet. 2018 Sep 22;392(10152):1036-1046. doi: 10.1016/S0140-6736(18)31924-X. Epub 2018 Aug 26. PMID 30158069
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Habib PJ, Green J, Butterfield RC, Kuntz GM, Murthy R, Kraemer DF, Percy RF, Miller AB, Strom JA. Association of cardiac events with coronary artery disease detected by 64-slice or greater coronary CT angiography: a systematic review and meta-analysis. Int J Cardiol. 2013 Oct 30;169(2):112-20. doi: 10.1016/j.ijcard.2013.08.096. Epub 2013 Sep 7. PMID 24090745
- [Background] Koo BK, Kang J, Park KW, Rhee TM, Yang HM, Won KB, Rha SW, Bae JW, Lee NH, Hur SH, Yoon J, Park TH, Kim BS, Lim SW, Cho YH, Jeon DW, Kim SH, Han JK, Shin ES, Kim HS; HOST-EXAM investigators. Aspirin versus clopidogrel for chronic maintenance monotherapy after percutaneous coronary intervention (HOST-EXAM): an investigator-initiated, prospective, randomised, open-label, multicentre trial. Lancet. 2021 Jun 26;397(10293):2487-2496. doi: 10.1016/S0140-6736(21)01063-1. Epub 2021 May 16. PMID 34010616
- [Background] Schlett CL, Banerji D, Siegel E, Bamberg F, Lehman SJ, Ferencik M, Brady TJ, Nagurney JT, Hoffmann U, Truong QA. Prognostic value of CT angiography for major adverse cardiac events in patients with acute chest pain from the emergency department: 2-year outcomes of the ROMICAT trial. JACC Cardiovasc Imaging. 2011 May;4(5):481-91. doi: 10.1016/j.jcmg.2010.12.008. PMID 21565735
- [Background] de Azevedo CF, Hadlich MS, Bezerra SG, Petriz JL, Alves RR, de Souza O, Rati M, Albuquerque DC, Moll J. Prognostic value of CT angiography in patients with inconclusive functional stress tests. JACC Cardiovasc Imaging. 2011 Jul;4(7):740-51. doi: 10.1016/j.jcmg.2011.02.017. PMID 21757164